CLINICAL TRIAL: NCT07044063
Title: Use of Diaphragm Ultrasound and Evaluation of Respiratory Parameters in Determining Weaning Success in Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ismail Yavuz Keles, Resident Doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: DLKTRH-ANS-IYK-01
Record Dates: First submitted 2025-04-09; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-04

CONDITIONS: Weaning Failure of Mechanical Ventilation; Diaphragm Ultrasonography; Geriatric
Keywords: diaphragm; ultrasound; geriatric; weaning; mechanical ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Weaning Success Group: Patients who are weaned from mechanical ventilation within 24 hours of diaphragmatic ultrasound measurements and didn't need mechanical ventilation again for at least 48 hours was placed in this group.
- Weaning Failure Group: Patients who are weaned from mechanical ventilation within 24 hours of diaphragmatic ultrasound measurements but needed mechanical ventilation support again within 48 hours after weaning was placed in this group.

SUMMARY:
This study aims to evaluate the effectiveness of ultrasound-based diaphragmatic measurements in predicting weaning success in patients aged 65 and older who are receiving mechanical ventilation. Additionally, it seeks to contribute to the clinical decision-making process by examining the relationship between these measurements and conventional weaning parameters.

DETAILED DESCRIPTION:
Weaning refers to the gradual reduction of mechanical ventilatory support. Approximately 40% of the time patients spend on mechanical ventilation is dedicated to the weaning process. Patients who fail the spontaneous breathing trial (SBT) or require reintubation within 48 hours after extubation are considered to have experienced weaning failure. Around 20-30% of patients receiving invasive mechanical ventilation are classified as difficult to wean.

In the geriatric population, the weaning process becomes even more challenging due to age-related changes such as decreased lung elasticity, reduced muscle mass, and diminished lung volumes. Although various scales have been developed to predict weaning success, their correlation with actual clinical outcomes remains uncertain.

The diaphragm is the primary muscle involved in active inspiration. Dysfunction of the diaphragm can lead to impaired cough reflex and respiratory failure. In recent years, ultrasonography (US) has been used to assess diaphragmatic thickness and movement through the right hemithorax during inspiration and expiration. From these measurements, parameters such as Diaphragm Thickness during inspiration and expiration (DTi and DTe), Diaphragm Thickening Fraction (DTF), and Diaphragm Excursion (DE) can be calculated. Several studies have investigated the association between these parameters and weaning success.

In this planned study, the investigators aim to evaluate the predictive value of ultrasound-derived diaphragmatic parameters (DTi, DTe, DTF, and DE) for weaning success in geriatric patients who are intubated and monitored in intensive care units. Additionally, investigators intend to assess the correlation between these parameters and other respiratory indicators.

The primary objective of this study is to examine the relationship between diaphragmatic parameters measured via ultrasonography within 24 hours prior to weaning and weaning outcomes in intubated ICU patients aged 65 years and older. The secondary objective is to compare the correlation of these parameters with other conventional respiratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Admitted to ICU
* Intubated and mechanically ventilated for at least 24 hours
* Clinically decided to wean from mechanical ventilation

Exclusion Criteria:

* Those who have mechanically ventilated for more than 14 days
* Those who have been tracheostomized
* Those with preexisting diaphragm or lung pathologies
* Those who had cardiothoracic surgery
* Those with muscular or musculoskeletal diseases
* Those with Glasgow Coma Scale lower than 10T without sedation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the intensive care unit of Kartal Dr. Lutfi Kirdar Training and Research Hospital who are 65 years or older and underwent mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Diaphragm Thickness Measurement | Within 24 hours prior to weaning from mechanical ventilation.
  Diaphragm thicknesses are measured with linear ultrasound probe at 8-10th intercostal space on anterior or middle axillary line using B-mode during inspiration and expiration.
Diaphragmatic Excursion Measurement | Within 24 hours prior to weaning from mechanical ventilation.
  Diaphragmatic excursion is measured with convex probe at midclavicular line just below costal arch using M-mode during respiratory cycle.
Diaphragm Thickening Fraction | Within 24 hours prior to weaning from mechanical ventilation.
  Diaphragmatic thickening fraction is calculated by taking the difference between diaphragm thickness at end-inspiration and diaphragm thickness at end-expiration, dividing it by the thickness at end-expiration, and multiplying by 100 to get a percentage.

SECONDARY OUTCOMES:
Arterial Blood Gas | Within 24 hours prior to weaning from mechanical ventilation.
  pH, Partial Pressure of Carbon Dioxide (mmHg) , Partial Pressure of Oxygen (mmHg), Oxygen Saturation(SaO2) values from arterial blood gas will be collected.
Oxygen Saturation | Within 24 hours prior to weaning from mechanical ventilation
  Peripheral Oxygen Saturation Percentage
Respiratory Rate (Breaths per Minute) | Within 24 hours prior to weaning from mechanical ventilation
  Respiratory rate per minute will be collected.
Rapid Shallow Breathing Index (Breath/Minute/L) | Within 24 hours prior to weaning from mechanical ventilation
  RSBI will be calculated by dividing respiratory rate per minute to tidal volume in liters.
Mechanical Ventilation Duration (Hours) | Within 24 hours prior to weaning from mechanical ventilation
  Mechanical ventilation duration prior to the weaning trial of the patients was recorded in hours.
PaO2/FiO2 (mmHg) | Within 24 hours prior to weaning from mechanical ventilation.
  PaO2 from arterial blood gas analysis was divided by fractional inspired oxygen to calculate this value.
Tidal Volume and Minute Ventilation (L) | Within 24 hours prior to weaning from mechanical ventilation.
  These values were collected from mechanical ventilator.
P0.1 (cmH2O) | Within 24 hours prior to weaning from mechanical ventilation.
  P0. 1 is the negative airway pressure generated by the patient during the first 0.1 s against an occluded airway. P0. 1 can be obtained non-invasively in most new generation mechanical ventilators through a simple maneuver.
Dynamic Compliance (mL/cmH2O) | Within 24 hours prior to weaning from mechanical ventilation.
  Dynamic compliance is measured by dividing the tidal volume, the average volume of air in one breath cycle, by the difference between the pressure of the lungs at full inspiration and full expiration. These values were collected from mechanical ventilator.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Kartal Dr. Lutfi Kirdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided